CLINICAL TRIAL: NCT00003387
Title: Concurrent Carboplatin, Paclitaxel, and Radiation Therapy Versus Induction Carboplatin and Paclitaxel Followed by Concurrent Carboplatin, Paclitaxel and Radiation Therapy for Patients With Unresectable Stage III Non-Small Cell Lung Cancer: A Phase III Trial
Brief Title: Carboplatin, Paclitaxel, and Radiation Therapy in Treating Patients With Stage III Non-small Cell Lung Cancer That Cannot Be Removed During Surgery
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Alliance for Clinical Trials in Oncology (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CALGB-39801; U10CA031946 (NIH); CLB-39801; CDR0000066383 (Registry Identifier: NCI Physician Data Query)
Record Dates: First submitted 1999-11-01; First posted 2003-11-26 (Estimated); Last update posted 2016-07-20 (Estimated); Status verified 2016-07

CONDITIONS: Lung Cancer
Keywords: stage III non-small cell lung cancer; squamous cell lung cancer; large cell lung cancer; adenocarcinoma of the lung
MeSH Terms: conditions — Lung Neoplasms; Carcinoma, Non-Small-Cell Lung; Adenocarcinoma of Lung | interventions — Carboplatin; Drug Therapy; Paclitaxel; Radiotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Chemo + radiation (Experimental)
  Interventions: Drug: carboplatin; Drug: chemotherapy; Drug: paclitaxel; Radiation: radiation therapy
- Induction chemo + chemo & radiation (Experimental)
  Interventions: Drug: carboplatin; Drug: chemotherapy; Drug: paclitaxel; Radiation: radiation therapy

INTERVENTIONS:
Drug: carboplatin
Drug: chemotherapy
Drug: paclitaxel
Radiation: radiation therapy

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die. Radiation therapy uses high-energy x-rays to damage tumor cells. It is not yet known whether giving chemotherapy before combined chemotherapy and radiation therapy is more effective than combined chemotherapy and radiation therapy alone in treating patients with non-small cell lung cancer.

PURPOSE: Randomized phase III trial to compare the effectiveness of carboplatin and paclitaxel followed by radiation therapy and chemotherapy with radiation therapy and chemotherapy alone in treating patients with stage III non-small cell lung cancer that cannot be removed during surgery.

DETAILED DESCRIPTION:
OBJECTIVES: I. Compare the effects of concurrent chemoradiotherapy utilizing carboplatin and paclitaxel with or without prior induction chemotherapy on overall response rate, disease-free survival, and overall survival in patients with unresectable stage III non-small cell lung cancer. II. Compare the effects of these treatments on locoregional vs distant failure in these patients. III. Compare the toxicity of these treatments in these patients.

OUTLINE: This is a randomized study. Patients are stratified by measurable vs evaluable disease. Patients are randomized to 1 of 2 treatment arms: Arm I (immediate concurrent chemoradiotherapy): Patients receive IV paclitaxel over 1 hour followed by IV carboplatin over 30 minutes on day 1, and radiation therapy to the chest 5 times a week beginning on day 1. Treatment repeats weekly for a total of 7 courses. Arm II (induction chemotherapy followed by delayed concurrent chemoradiotherapy): Patients receive IV paclitaxel over 3 hours followed by IV carboplatin over 30 minutes; treatment repeats every 3 weeks for 2 courses. Patients then receive 7 courses of concurrent chemoradiotherapy as in Arm I. Total treatment time is 13 weeks. Patients are followed every 2 months for 2 years, then every 4 months for the next 2 years, then annually thereafter.

PROJECTED ACCRUAL: A total of 360 patients will be accrued for this study within 3 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS: Histologically or cytologically confirmed non-small cell lung cancer, including: Squamous cell carcinoma Adenocarcinoma (including bronchoalveolar cell) Large cell anaplastic carcinoma (including giant and clear cell carcinomas) Inoperable or unresectable stage IIIA or IIIB disease of the following stage groupings: T1 N2 M0 or T2 N2 M0 T3 N2 M0 and T4 N0-2 M0 eligible if staging is based on closeness to the carina or invasion of the mediastinum or chest wall Patients with contralateral mediastinal disease (N3) or tumors adjacent to but not invading a vertebral body are eligible if all gross disease can be encompassed in the study radiation boost field Patients with a transudate, cytologically negative, nonbloody pleural effusion are eligible if the tumor can be encompassed within a reasonable field of radiotherapy Measurable or evaluable disease

PATIENT CHARACTERISTICS: Age: 18 and over Performance status: CALBG 0-1 Life expectancy: Not specified Hematopoietic: Platelet count at least 100,000/mm3 Absolute granulocyte count at least 1,500/mm3 Hepatic: Bilirubin less than 1.5 mg/dL AST less than 2 times upper limit of normal Renal: Creatinine clearance at least 20 mL/min Other: Not pregnant or nursing Effective contraception required of fertile patients No active second malignancy except nonmelanomatous skin cancer

PRIOR CONCURRENT THERAPY: Biologic therapy: Not specified Chemotherapy: No prior chemotherapy No other concurrent chemotherapy Endocrine therapy: No concurrent hormones except for steroids administered for adrenal failure or septic shock, or hormones administered for non-disease-related conditions (e.g., insulin for diabetes) Glucocorticosteroids permitted as antiemetics Radiotherapy: No prior radiotherapy Surgery: At least 2 weeks since exploratory thoracotomy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 366 (Actual)
Dates: Start 1998-07; Primary Completion 2007-05 (Actual); Study Completion 2009-04 (Actual)

PRIMARY OUTCOMES:
overall response rate | Up to 5 years
overall survival | Up to 5 years
disease-free survival | Up to 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Everett E. Vokes, MD, Study Chair — University of Chicago
Locations (47):
- United States (47):
  - Veterans Affairs Medical Center - Birmingham, Birmingham, Alabama
  - University of California San Diego Cancer Center, La Jolla, California
  - Veterans Affairs Medical Center - San Francisco, San Francisco, California
  - UCSF Cancer Center and Cancer Research Institute, San Francisco, California
  - CCOP - Christiana Care Health Services, Wilmington, Delaware
  - Howard University Cancer Center, Washington D.C., District of Columbia
  - Walter Reed Army Medical Center, Washington D.C., District of Columbia
  - CCOP - Mount Sinai Medical Center, Miami Beach, Florida
  - University of Illinois at Chicago Health Sciences Center, Chicago, Illinois
  - Veterans Affairs Medical Center - Chicago (Westside Hospital), Chicago, Illinois
  - University of Chicago Cancer Research Center, Chicago, Illinois
  - Hematology Oncology Associates of the Quad Cities, Bettendorf, Iowa
  - Holden Comprehensive Cancer Center at The University of Iowa, Iowa City, Iowa
  - Veterans Affairs Medical Center - Togus, Togus, Maine
  - Marlene & Stewart Greenebaum Cancer Center, University of Maryland, Baltimore, Maryland
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - University of Massachusetts Memorial Medical Center, Worcester, Massachusetts
  - Veterans Affairs Medical Center - Minneapolis, Minneapolis, Minnesota
  - Veterans Affairs Medical Center - Columbia (Truman Memorial), Columbia, Missouri
  - Ellis Fischel Cancer Center - Columbia, Columbia, Missouri
  - Barnes-Jewish Hospital, St Louis, Missouri
  - University of Nebraska Medical Center, Omaha, Nebraska
  - CCOP - Southern Nevada Cancer Research Foundation, Las Vegas, Nevada
  - Norris Cotton Cancer Center, Lebanon, New Hampshire
  - Cooper Cancer Institute, Camden, New Jersey
  - Veterans Affairs Medical Center - Buffalo, Buffalo, New York
  - Roswell Park Cancer Institute, Buffalo, New York
  - CCOP - North Shore University Hospital, Manhasset, New York
  - North Shore University Hospital, Manhasset, New York
  - Memorial Sloan-Kettering Cancer Center, New York, New York
  - New York Presbyterian Hospital - Cornell Campus, New York, New York
  - Mount Sinai Medical Center, NY, New York, New York
  - State University of New York - Upstate Medical University, Syracuse, New York
  - Veterans Affairs Medical Center - Syracuse, Syracuse, New York
  - CCOP - Syracuse Hematology-Oncology Associates of Central New York, P.C., Syracuse, New York
  - Lineberger Comprehensive Cancer Center, UNC, Chapel Hill, North Carolina
  - Veterans Affairs Medical Center - Durham, Durham, North Carolina
  - Duke Comprehensive Cancer Center, Durham, North Carolina
  - CCOP - Southeast Cancer Control Consortium, Winston-Salem, North Carolina
  - Comprehensive Cancer Center at Wake Forest University, Winston-Salem, North Carolina
  - Rhode Island Hospital, Providence, Rhode Island
  - Medical University of South Carolina, Charleston, South Carolina
  - University of Tennessee, Memphis Cancer Center, Memphis, Tennessee
  - Veterans Affairs Medical Center - Memphis, Memphis, Tennessee
  - Veterans Affairs Medical Center - White River Junction, White River Junction, Vermont
  - Veterans Affairs Medical Center - Richmond, Richmond, Virginia
  - MBCCOP - Massey Cancer Center, Richmond, Virginia

REFERENCES:
- [Result] Stinchcombe TE, Hodgson L, Herndon JE 2nd, Kelley MJ, Cicchetti MG, Ramnath N, Niell HB, Atkins JN, Akerley W, Green MR, Vokes EE; Cancer and Leukemia Group B. Treatment outcomes of different prognostic groups of patients on cancer and leukemia group B trial 39801: induction chemotherapy followed by chemoradiotherapy compared with chemoradiotherapy alone for unresectable stage III non-small cell lung cancer. J Thorac Oncol. 2009 Sep;4(9):1117-25. doi: 10.1097/JTO.0b013e3181b27b33. PMID 19652624
- [Result] Vokes EE, Herndon JE 2nd, Kelley MJ, Cicchetti MG, Ramnath N, Neill H, Atkins JN, Watson DM, Akerley W, Green MR; Cancer and Leukemia Group B. Induction chemotherapy followed by chemoradiotherapy compared with chemoradiotherapy alone for regionally advanced unresectable stage III Non-small-cell lung cancer: Cancer and Leukemia Group B. J Clin Oncol. 2007 May 1;25(13):1698-704. doi: 10.1200/JCO.2006.07.3569. Epub 2007 Apr 2. PMID 17404369